CLINICAL TRIAL: NCT06937957
Title: A Phase I Study to Investigate the Safety, Pharmacokinetics, Immunogenicity and Efficacy of BR111 for Injection in Patients With Advanced Malignancies
Brief Title: A Study of BR111 in Patients With Advanced Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BioRay Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR111-101
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Advanced Malignancies
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Does escalation (Experimental)
  Interventions: Drug: BR111 for Injection

INTERVENTIONS:
Drug: BR111 for Injection — BR111-101 for injection will be administered by intravenous drip, disease progression, pregnancy, withdrawal of informed consent, death, study discontinuation or withdrawal from the study. The dose of each administration will be calculated based on the weight measured prior to such administration. The dosing regimen (dosing frequency and interval) for subsequent study may be adjusted based on prior data. The intravenous drip should last for ≥ 90 min for the first dose and may be adjusted to ≥ 30 min for subsequent doses if the first dose is tolerable.
Drug: BR111 for Injection — BR111-101 for injection will be administered via intravenous drip at a fixed frequency and cycle until intolerable toxicity, disease progression, pregnancy, withdrawal of informed consent, death, study discontinuation, or withdrawal from the study occurs. The dose for each administration will be calculated based on the body weight measured prior to administration. The dosing regimen (dosing frequency and interval) for subsequent studies may be adjusted based on prior data. The intravenous drip duration should be ≥ 90 minutes for the first dose and may be adjusted to ≥ 30 minutes for subsequent doses if the first dose is well tolerated.

SUMMARY:
This is a Phase I, multicenter, open-label, single-arm and first-in-human clinical study of BR111-101 for injection. The study objectives are to evaluate the safety, tolerability, pharmacokinetic profile, anti-tumor activity and immunogenicity of BR111-101 for injection in patients with advanced malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to provide written informed consent for the study;
2. Age ≥ 18 years, male or female; Patients with solid tumors: Patients with histopathologically confirmed advanced solid tumors who are not amenable to surgical resection who have failed standard therapy (i.e., existing therapies with known clinical benefit) (disease progression during or after treatment) or who cannot tolerate standard therapy and are unable to obtain or refuse or have no standard therapy.

   Patients with lymphoma: Patients with histopathologically confirmed relapsed/refractory B-cell lymphoma who meet the 2016 WHO classification criteria and are indicated for treatment and currently have no other standard treatment as judged by the investigator.
3. All patients are required to provide tumor samples for biomarker analysis at screening.
4. ECOG score 0 to 1 .
5. Life expectancy ≥ 3 months.
6. Phase Ia dose Escalation: Patients with solid tumors or lymphoma have at least one evaluable lesion at baseline (ie, no measurable lesions) according to RECIST v1.1 or Lugano 2014 criteria; Phase Ia Safety Expansion and Phase Ib: Patients with at least 1 measurable lesion at baseline according to RECISTv1.1 and Lugano 2014 criteria. Lesions previously treated with radiotherapy or intervention should not be considered target lesions unless there is unequivocal progression.
7. Adequate organ and bone marrow function ；
8. Female patients of childbearing potential (defined as those who are not surgically sterile with hysterectomy and/or bilateral oophorectomy and are not postmenopausal, defined as having amenorrhea ≥ 12 months) must have a negative pregnancy test at entry into this study and must be non-lactating; female patients of childbearing potential or male patients with sexual partners of childbearing potential are willing to use appropriate effective contraceptive measures such as abstinence and double-barrier methods (e.g., condom plus diaphragm), oral contraceptives, and placement of an intrauterine device during the study and for 6 months after the last investigational product.
9. Able to understand trial requirements and willing and able to comply with trial and follow-up procedures.

Exclusion Criteria:

Patients will not be eligible to participate in the study if they meet any of the following exclusion criteria:

1. Has unresolved toxicities from previous anticancer therapy, defined as toxicities not yet resolved to NCI CTCAE 5.0, Grade ≤1 or baseline（except for alopecia, pigmentation, or other toxicities judged by the investigator to have no safety risk）；
2. Known history of allergy or delayed allergic reactions to BR111 for Injection and its components and considered severe by the investigator;
3. Prior use of eribulin, or the treatments or clinical trials based on eribulin , or prior use of drugs or clinical trials targeting ROR1;
4. Primary central nervous system malignancy or invasion of the central nervous system (Patients with CNS invasion may be considered for enrollment if they are untreated but asymptomatic, or with CNS metastases that have been radiologically documented to be progression-free for at least 4 weeks and require no treatment for at least 4 weeks). ;
5. Patients with bacterial, viral, fungal, mycobacterial, parasitic or other infections within 14 days before the first dose and requiring intravenous infusion therapy (except for neoplastic fever);
6. Patients with a history of (non-infectious) interstitial lung disease/pneumonia requiring steroid therapy, or current interstitial lung disease/non-infectious pneumonia, or suspected interstitial lung disease/non-infectious pneumonia that cannot be excluded by imaging at screening; radiation pneumonitis patients without clinical symptoms after 3 months of radiotherapy can be enrolled;
7. Advanced malignant tumor complications resulting in quiescent dyspnea or current need for continuous oxygen therapy;
8. Patients with moderate to severe lung diseases that have clinically significant impact on lung function, including but not limited to pulmonary embolism, severe asthma, severe chronic obstructive pulmonary disease, idiopathic pulmonary fibrosis, or previous pneumonectomy within 3 months before enrollment;
9. Peripheral neuropathy of Grade ≥ 2 (refer to NCI CTCAE 5.0) ;
10. Accompanied by severe cardiovascular and cerebrovascular diseases or other serious organic diseases, including but not limited to:

    * Stroke, intracranial hemorrhage, unstable angina pectoris, congestive heart failure (NYHA Class III-IV), myocardial infarction, severe arrhythmia (such as sustained ventricular tachycardia, ventricular fibrillation), congenital long QT syndrome, torsades de pointes, etc. within 6 months prior to the first dose;
    * Left ventricular ejection fraction LVEF < 50% by echocardiography (ECHO) or multiple-gated acquisition (MUGA) scan;
    * Mean corrected QT interval prolongation > 470 ms in 3 consecutive ECGs during the screening period, and QT interval correction (QTcF) is performed using the F ridercia formula;
    * Grade ≥3 hypertension that cannot be stably controlled (refer to NCI CTCAE 5.0);
    * Known inherited or acquired bleeding disorders or significant coagulation abnormalities (e.g., disseminated intravascular coagulation (DIC), autoimmune anemia, etc.)
11. Complete intestinal obstruction before the first dose, or pericardial effusion with clinical symptoms requiring drainage, or pleural and peritoneal effusion, or skin lesions that are difficult to heal, recurrent episodes of any cause, and/or nonhealing ulcers (except for cancerous ulceration);
12. Patients with previous or suspected serious skin conditions prior to first dose, including but not limited to bullous or exfoliative dermatitis, erythema multiforme, toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome (SJS), and drug reaction with eosinophilia and systemic symptoms (DRESS);
13. Patients with immunodeficiency or active autoimmune diseases (except those with immune-related adverse reactions caused by previous application of immune checkpoint inhibitors that are relieved or stabilized at grade 1 after treatment) or requiring systemic steroid therapy. For patients with solid tumors: systemic corticosteroids at doses > 10 mg/day prednisone or equivalent hormone for more than 1 week within 14 days prior to first dose; for patients with lymphoma: systemic corticosteroids at doses > 20 mg/day prednisone or equivalent hormone for more than 1 week within 14 days prior to first dose ;
14. Any other malignancy within 3 years (except basal cell carcinoma of the skin that has been radically treated and has not recurred, squamous cell carcinoma of the skin, superficial bladder cancer, localized prostate cancer, cervical cancer in situ, ductal carcinoma in situ of the breast, and malignancies that have been cured (CR) within 2 years prior to the first dose and judged by the investigator to be in stable disease status with minimal risk of recurrence);
15. HIV virus test positive; syphilis infection requiring systemic treatment; HCVAb positive with HCV RNA titer above the upper limit of normal detected at the same time; Patients with solid tumors: HBsAg positive with HBV DNA ≥ 500 IU/mL at the same time; Patients with lymphoma: HBsAg positive or HBcAb positive, simultaneous HBV DNA ≥ 500 IU/mL;
16. Participated in other clinical trial treatment within 4 weeks prior to the first dose (i.e., within 4 weeks from the last clinical trial drug/device treatment); Note: If the human half-life of the investigational product is clearly known, there should be an interval of at least 4 weeks or 5 half-lives (whichever is shorter) between the patient's previous clinical trial medication and the first dose of BR111;
17. Major surgery or serious trauma within 4 weeks prior to the first dose that has not fully recovered or surgery is expected during the trial ;
18. Received anti-tumor therapy such as radiotherapy and targeted therapy within 4 weeks prior to the first dose of study drug, as well as the following:

    Received nitrosoureas (e.g., carmustine, romosustine, etc.) or mitomycin C within 6 weeks before the first dose; palliative radiotherapy for bone metastases or local radiotherapy for pain relief within 2 weeks before the first dose; chemotherapy, small molecule targeted drugs, endocrine therapy, or fluorouracil within 2 weeks before the first dose, but patients with prostate cancer are allowed to continue luteinizing hormone-releasing hormone (LHRH) agonist/antagonist therapy during the study; and traditional Chinese medicines or modern traditional Chinese medicine preparations with anti-tumor indications within 2 weeks before the first dose;
19. Previous allogeneic hematopoietic stem cell transplantation or solid organ transplantation or autologous hematopoietic stem cell transplantation less than 3 months before the first dose or CAR-T cell therapy less than 3 months before the first dose;
20. Any mental or cognitive impairment that may limit their understanding and execution of the informed consent form;
21. Other serious, uncontrolled concomitant diseases that may affect protocol compliance or interfere with the results or other serious or uncontrollable disease conditions that, in the opinion of the investigator, may pose a risk to the patient by participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2027-10-09 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of BR111 if any (for dose escalation part) | About 9 months
  Participants will receive BR111 for injection once every three weeks. The MTD will be determined by the number of participants who experience a dose limiting toxicity (DLT).
Recommended Phase 2 Dose(RP2D) of BR111 (for dose escalation part) | About 9 months
  The selection of RP2D will be based on consideration of overall safety information together with available pharmacokinetic, pharmacodynamic, and efficacy data. The RP2D may be the MTD or may be a lower dose within the tolerable dose range.

SECONDARY OUTCOMES:
Incidence of anti-drug antibodies (ADA) | Until 30 days since the last dose of investigational product or until initiation of a new anti-cancer treatment, whichever occurs first
Incidence of Neutralizing antibodies (Nab) | Until 30 days since the last dose of investigational product or until initiation of a new anti-cancer treatment, whichever occurs first
Concentration of BR111 total antibody, prodrug and the free cytotoxin | Until 30 days since the last dose of investigational product or until initiation of a new anti-cancer treatment, whichever occurs first
objective response rate（ORR） | Until 30 days since the last dose of investigational product or until initiation of a new anti-cancer treatment, whichever occurs first
  Objective Response Rate is defined as the percentage of patients with a complete response (CR) or partial response (PR)

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Cancer, Shanghai, Pudong New Area, China

IPD SHARING:
Plan to Share IPD: No